CLINICAL TRIAL: NCT04398849
Title: Immunisation for Adolescents Against Serious Communicable Diseases
Brief Title: Immunisation for Adolescents Against Serious Communicable Diseases (B Part of it NT)
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Adelaide (Other)
Collaborators: The University of New South Wales (Other); Menzies School of Health Research (Other); University of Sydney (Other); The University of Western Australia (Other); Northern Territory Government of Australia (Other Government); SA Health (Other); The University of Queensland (Other)
Responsible Party: Principal Investigator, Helen Marshall, Professor, University of Adelaide
Other Study IDs: Menzies HREC/2019-3507-V1.7
Record Dates: First submitted 2020-05-18; First posted 2020-05-21 (Actual); Last update posted 2023-03-09 (Actual); Status verified 2023-03

CONDITIONS: Gonorrhea; Meningococcal Disease
MeSH Terms: conditions — Gonorrhea; Meningococcal Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Oropharyngeal swab specimens
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- 14-19 year olds residing in the Northern Territory: All consenting 14-19 year olds residing in the Northern Territory in 2020-2021
  Interventions: Biological: Licenced 4CMenB Vaccine

INTERVENTIONS:
Biological: Licenced 4CMenB Vaccine — Two doses (0.5 mL each) of Bexsero ® vaccine at least 2 months apart to be given to consenting 14-19 year olds

SUMMARY:
This study aims to implement a targeted 4CMenB immunisation program in young people aged 14-19 years in the Northern Territory (NT). As part of the NT program consenting 14-19 year olds will receive 2 doses of the licensed 4CMenB vaccine. An oropharyngeal swab will be collected on the same day as the first dose of the vaccine and 12 months later to assess carriage of Neisseria meningitidis. The first swab will assess baseline carriage prevalence among 14-19 year olds in the NT. The swab taken 12 months later will provide data on the change in carriage that may occur after implementation of the immunisation program. Emerging evidence suggests that the 4CMenB vaccine may be protective against gonorrhea. Therefore, vaccine effect (impact and effectiveness) against both invasive meningococcal disease (IMD) and gonorrhea in the NT will be assessed using data from the above study comparing notifications between vaccinated and unvaccinated as well as comparing pre and post implementation periods.

DETAILED DESCRIPTION:
Meningococcal disease and gonorrhea cause severe morbidity in Australian adolescents, particularly among Aboriginal People. The two diseases are caused by bacteria that are genetically related, but very different in their patterns of transmission and pathogenesis. Bacterial meningitis and sepsis from Neisseria meningitidis (often called meningococcus) can have severe outcomes including long-term disability, arising from neurological deficits and from necrotic skin and gangrene of the limbs requiring amputations. The case fatality rate is ~10%. A multicomponent meningococcal B (4CMenB) vaccine (Bexsero®) is approved and licensed for use against MenB disease in Australia but not funded on the National Immunisation Program (NIP) due to failure to meet cost effectiveness criteria. New emerging data suggest 4CMenB may also protect against gonococcal infection, a sexually transmissible infection (STI) which can infect the urethra, cervix, rectum, conjunctiva, and throat. If left untreated, gonorrhoea can lead to pelvic inflammatory disease, tubal scarring and ultimately infertility in females, and swelling and scarring in the epididymis or testicles in males. In the NT, notification rates for gonorrhoea in 15-19 year olds range from 1924/100,000 to 17,022/100,000 in Aboriginal young people and from 106/100,000 to 1081/100,000 in non-Aboriginal young people over different areas of The Territory (averaged over 2014-2018). At present there is no vaccine against gonorrhoea. Emerging evidence shows that the 4CMenB vaccine may have some protection against gonorrhoea due to genetic similarities that exist between the two organisms that cause meningitis and gonorrhoea. If the effectiveness of the 4CMenB vaccine against gonorrhoea can be demonstrated at a population level it would have substantial health benefits to be gained world-wide, but particularly for Aboriginal People.

Consenting 14-19 year olds will be asked to complete a 1-2 page questionnaire to collect information on risk factors for meningococcal disease and meningococcal carriage. A throat swab will be obtained and the first dose of the 4CMenB vaccine will be administered. Two-three months after the first dose, participants will receive the second dose of the 4CMenB vaccine. One year after the first dose, the participants will be asked to come for the third visit, where they will be asked to complete the same questionnaire that was completed during visit one and a throat swab taken. Throat swabs will be tested to detect the meningococcus bacteria which is carried in the throat of around 10% of people. Research in South Australia has shown double the rates of carriage in Aboriginal People compared to non-Aboriginal People.

The effectiveness of the 4CMenB vaccine against meningococcal carriage, invasive meningococcal disease and gonorrhoea will be evaluated using results of meningococcal carriage and routine surveillance data on IMD and gonorrhoea obtained from the Centre for Disease Control (CDC), the data custodian for notifiable diseases in the NT. The evaluations will include comparisons between vaccinated vs unvaccinated and number of notifications in post vs pre study implementation periods. The data on IMD and gonorrhoea notifications in the NT will be obtained from the Communicable Disease Control in the NT. The main methodological approaches involve an Interrupted Time Series regression model, screening approaches, and case-control analyses with different sets of controls to estimate vaccine impact and effectiveness

ELIGIBILITY:
Inclusion Criteria:

All consenting 14-19 year olds residing in the Northern Territory in 2020-2021

Exclusion Criteria:

* Anaphylaxis following any component of Bexsero® vaccine
* Previous receipt of MenB vaccine (Bexsero® (Previous receipt of MenNZBTM is allowed).
* Known pregnancy
* Clinical conditions representing a contraindication to intramuscular vaccination and venipuncture
* Any clinical condition that, in the opinion of the investigator, might pose additional risk to the subject due to participation in the study

Ages: 14 Years to 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: All consenting 14-19-year-olds residing in the Northern Territory who do not have any of the above exclusion criteria
Sampling Method: Non-Probability Sample
Enrollment: 7100 (Estimated)
Dates: Start 2021-03-04 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
1. 4CMenB vaccination status in the population with gonorrhoea compared to randomly selected Chlamydia controls (Case-control) | 3 years
  Vaccination status among 15-19 year olds diagnosed with gonorrhoea compared to vaccination status of 15 - 19 year olds diagnosed with Chlamydia
Effect of 4CMenB vaccine on carriage of all N.meningitidis | 12 months
  Prevalence of all N. meningitidis in the pharynx among 14-19 year olds as measured by PCR at baseline compared to 12 months

SECONDARY OUTCOMES:
4CMenB vaccination status in the population with gonorrhoea compared to randomly selected controls from the Australian Immunisation Register (Case-control) | 3 years
  4CMenB vaccination status among 15-19 year olds diagnosed with gonorrhoea compared to controls from the Australian Immunisation register
4CMenB vaccination status in the population with gonorrhoea compared to the general population (Screening method) | 3 years
  4CMenB vaccination status among 15-19 year olds diagnosed with gonorrhoea compared to the general population
All laboratory confirmed notifications of gonorrhoea in the six years preceding 4CMenB vaccination compared to three years post vaccination (Interrupted time series analysis) | 7 years
  Laboratory confirmed notifications of gonorrhoea in years preceding 4CMenB vaccination compared to post vaccination
All laboratory confirmed notifications of gonorrhoea in 15-19 year olds in the vaccinated population compared to the unvaccinated population | 3 years
  Gonorrhoea notifications in vaccinated vs unvaccinated
All laboratory confirmed notifications of gonorrhoea in the vaccinated population compared to the unvaccinated population stratified by gender | 3 years
  Gonorrhoea notifications in vaccinated vs unvaccinated (stratified by gender)
All laboratory confirmed notifications of gonorrhoea in the vaccinated population compared to the unvaccinated population stratified by geographical location (regional/remote/very remote) | 3 years
  Gonorrhoea notifications in vaccinated vs unvaccinated stratified by location
Effect of 4CMenB vaccine on carriage of all disease causing N.meningitidis | 12 months
  Prevalence of all disease-causing genogroup of N. meningitidis (A, B, C, E, X, W, Y) by PCR at baseline and at 12 months
Effect of 4CMenB vaccine on carriage of each disease causing N.meningitidis | 12 months
  Prevalence of each disease-causing genogroup of N. meningitidis (A, B, C, E, X, W, Y) by PCR at baseline and at 12 months
Effect of 4CMenB vaccine on carriage of all non-groupable N.meningitidis | 12 months
  Prevalence of all non groupable N. meningitidis at baseline and at 12 months
Effect of 4CMenB vaccine on acquisition of all N. meningitidis | 12 months
  Acquisition of all N. meningitidis (negative at baseline, positive at 12-month follow-up) as measured by PCR
Effect of 4CMenB impact on Group B IMD (Interrupted time series) | 3 years
  Notifications of group B IMD (invasive meningococcal disease) in the 4CMenB vaccinated population compared to the unvaccinated population and in years preceding 4CMenB vaccination compared to post vaccination (Interrupted time series analysis).
Effect of 4CMenB effectiveness on Group B IMD (screening method) | 3 years
  4CMenB vaccination status in the population with IMD, compared to the general population (Screening method) and compared to randomly selected controls (Case-control method).
Effect of 4CMenB effectiveness on Group B IMD (case-control method) | 3 years
  4CMenB vaccination status in the population with IMD, compared to the general population (Screening method) and compared to randomly selected controls (Case-control method).
Risk factors for gonorrhoea | 12 months
  Risk factors associated with gonorrhoea in 15-19 year olds
Risk factors for carriage of all N.meningitidis | 12 months
  Risk factors associated with carriage of all genogroups of N. meningitidis in 14 -19 year olds at baseline and 12 months
Risk for carriage of disease causing genogroups of N.meningitidis | 12 months
  Risk factors associated with carriage of disease-causing genogroups of N. meningitidis (A, B, C, E, W, X, Y) in 14 -19 year olds at baseline and 12 months
Cost effectiveness of the 4CMenB vaccine | 3 years
  Cost of meningococcal disease (acute care and management of sequelae up to one year) and cost of treatment of gonorrhoea compared to cost of 4CMenB vaccine

OTHER OUTCOMES:
Whole genome sequencing of all carriage isolates | 12 months
  Description of whole genome sequencing of all carriage isolates
Whole genome sequencing of all disease causing carriage isolates | 12 months
  Description of Whole genome sequencing of all disease causing carriage isolates
Awareness of STIs and STI testing among young adults | 12 months
  Proportion of 14 -19 year olds who undergo STI testing after implementation of the program compared to 12 months pre implementation

CONTACTS AND LOCATIONS:
Locations (1):
- Northern Territory, Central Australia, Australia

IPD SHARING:
Plan to Share IPD: Yes
De-identified, individual participant data underlying published results will be available
Supporting Information: Study Protocol, SAP
Time Frame: We estimate the data will be available from the start of 2025 for approximately 12 months
Access Criteria: IPD will be made available on a case-by-case basis at the discretion of the International Scientific Advisory Committee and The NT Department of Health and Menzies School of Health Research and the Central Australian HREC. IPD data will only be available to achieve the aims in the approved proposal

REFERENCES:
- [Derived] Marshall HS, Andraweera PH, Ward J, Kaldor J, Andrews R, Macartney K, Richmond P, Krause V, Koehler A, Whiley D, Giles L, Webby R, D'Antoine H, Karnon J, Baird R, Lawrence A, Petousis-Harris H, De Wals P, Greenwood-Smith B, Binks M, Whop L. An Observational Study to Assess the Effectiveness of 4CMenB against Meningococcal Disease and Carriage and Gonorrhea in Adolescents in the Northern Territory, Australia-Study Protocol. Vaccines (Basel). 2022 Feb 16;10(2):309. doi: 10.3390/vaccines10020309. PMID 35214767